CLINICAL TRIAL: NCT03951363
Title: Using Digital Health to Improve Diet and Exercise Adherence for Chronic Kidney Disease Management
Brief Title: iControl Chronic Kidney Disease
Acronym: iControl CKD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to COVID-19
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00101993
Record Dates: First submitted 2019-05-14; First posted 2019-05-15 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qualitative Interview (No Intervention): Interviews: The investigators will enroll at least 10 adults 18 years or older with CKD (self-report).
- Pilot Testing (Other): Pilot Study: The investigators will enroll 30 adults at least 18 years old with mild to moderate CKD (documented estimated glomerular filtration rate (eGFR) ≥60 ml/min/1.73m2 plus albuminuria or eGFR 45-59 ml/min/1.73m2) who also have diabetes and/or hypertension.
  Interventions: Behavioral: interactive Obesity Treatment Approach (iOTA)

INTERVENTIONS:
Behavioral: interactive Obesity Treatment Approach (iOTA) — The investigators will adapt an evidence-based digital health intervention to promote adherence to nationally recommended diet and physical activity guidelines for patients with chronic kidney disease. The intervention includes goal assignment, goal tracking, and skills training messages.
  Arms: Pilot Testing

SUMMARY:
The proposed study is responsive to the call for obtaining enhanced preliminary data for an external grant resubmission. The goal is to demonstrate a novel approach using digital health tools to help preserve kidney function. The investigators aim to adapt a previous behavioral intervention and conduct formative testing among patients with CKD. Specifically, the investigators will:

Aim 1: Modify an existing technology platform to build the iControl CKD system and adapt intervention content to reflect behavioral guidelines for patients with mild to moderate CKD.

Aim 2: Conduct qualitative interviews and user testing among patients with CKD to obtain feedback on the design of the intervention.

Aim 3: Conduct a prospective cohort feasibility trial to assess the feasibility and initial acceptability of the iControl CKD intervention.

ELIGIBILITY:
Inclusion criteria:

Qualitative interview:

* Age 18 or older
* Diagnosed with CKD (self-report)
* Proficient in English

Inclusion criteria:

Pilot Groups:

* Age 18 or older
* Diagnosed with mild to moderate CKD (documented eGFR ≥60 ml/min/1.73m2 plus albuminuria or eGFR 45-59 ml/min/1.73m2 )
* Diagnosed with diabetes and/or hypertension
* Proficient in English
* Access to a test-enabled mobile phone
* Willing to receive and send multiple text messages in a week

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Proportion of participants responding to Interactive Voice Response (IVR) calls or text tracking prompts | Approximately 1 Month
  Engagement with the intervention will be measured by calculating the proportion of participants responding to IVR calls or text tracking prompts over 1 month

SECONDARY OUTCOMES:
Change in CKD diet adherence as measured through consumption of CKD-specific nutrients (i.e. sodium, protein, potassium, and phosphorus) | Approximately 1 Month
  Analysis of 24-hour dietary recalls (1 weekday and 1 weekend day) at the beginning and end of the 1 month period
Change in physical activity minutes | Approximately 1 month
  Self-reported physical activity will be measured via the Paffenbarger Exercise Habits Questionnaire pre- and post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Dori Steinberg, PhD, RD, Principal Investigator — Duke University
Locations (1):
- Duke Global Digital Health Science Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No